CLINICAL TRIAL: NCT04813705
Title: A Multicenter Phase II Study of 18F-FDG PET/CT Guided Reduced-dose Radiotherapy for Nasopharyngeal Carcinoma
Brief Title: 18F-FDG PET/CT Guided Reduced-dose Radiotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Collaborators: Taizhou Enze Medical Center Group (Other); Taizhou Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Haihua Yang, Head of Department of Radiation Oncology, Taizhou Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRR-202103
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Off-Label Use; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced dose group (Experimental): The patients achieving CMR and more than 70% PMR at 25th fraction will receive reduced-dose radiotherapy for 30 fractions.
  Interventions: Radiation: Reduced dose; Drug: Chemotherapy
- Conventional dose group (Active Comparator): The patients who do not achieve CMR or 70% PMR at 25th fraction will receive conventional dose radiotherapy for 33 fractions.
  Interventions: Radiation: Conventional dose; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Reduced dose — The patients with CMR and more than 70% PMR at 25th fraction will receive reduced-dose radiotherapy for 30 fractions.
  Arms: Reduced dose group
Radiation: Conventional dose — The patients who do not achieve CMR or 70% PMR at 25th fraction will receive conventional dose radiotherapy for 33 fractions.
  Arms: Conventional dose group
Drug: Chemotherapy — The patients with stage II will receive concurrent cisplatin during Intensity modulated radiotherapy (IMRT), and stage III-IVA patients will receive platinum based induction chemotherapy every 21 days for at least two cycles followed by concurrent cisplatin during IMRT.

SUMMARY:
The purpose of this study is to explore whether 18F-FDG PET/CT guided reduced-dose radiotherapy would maintain survival outcomes in nasopharyngeal carcinoma (NPC) patients.

DETAILED DESCRIPTION:
Enrolled patients with complete metabolic response (CMR) and more than 70% partial metabolic response (PMR) according to PERCIST criteria at the 25th fraction will receive intensity modulated radiation therapy (IMRT) of reduced-dose (prescribed dose, 63.6 Gy, 2.12 Gy per fractions, 30 fractions), for those who with ≤70% PMR will receive conventional dose (prescribed dose, 70Gy, 2.12 Gy per fractions, 33 fractions).

ELIGIBILITY:
Inclusion Criteria:

1. Pathology confirmed nasopharyngeal squamous cell carcinoma.
2. Stage I-IVA（8thAJCC/UICC staging system).
3. Aged 18-80 years.
4. KPS≥70.
5. Have measurable lesions on 18F-FDG PET/CT before treatment.
6. HGB≥90 g/L，ANC≥1.5×109 /L，PLT≥80×109 /L.
7. ALT,AST<2.5 fold of ULN；TBIL<2.0×ULN.
8. CCR≥60ml/min or Cr<1.5×ULN.
9. Signed informed consent.
10. Have follow up condition.

Exclusion Criteria:

1. Past malignancies history (except for stage I non-melanoma skin cancer or cervical carcinoma in situ).
2. Age <18 or >80years.
3. Pregnancy or lactation.
4. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
5. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
6. With sever infection and internal disease.
7. Major organ dysfunction, such as decompensated cardiopulmonary, kidney, liver failure, cannot tolerate surgical treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Local-regional recurrence free survival (LRFS) | 5 years
  The LRFS is evaluated and calculated from the date of initiation of treatment until the day of first locoregional relapse or until the date of the last follow-up visit.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  The OS was defined as the duration from the date of of initiation of treatment to the date of death from any cause or censored at the date of the last follow-up.
Progression free survival (PFS) | 5 years
  Progress-free survival is calculated from the date of initiation of treatment to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.
Distant metastasis-free survival (DMFS) | 5 years
  The DMFS is evaluated and calculated from the date of initiation treatment until the day of first distant metastases or until the date of the last follow-up visit.
Incidence of treatment related acute complications | up to 3 months
  treatment-related adverse events will be assessed by NCI-CTC5.0 criteria and RTOG/EORTC criteria.
Incidence of treatment related late complications | up to 5 years
  treatment-related adverse events will be assessed by NCI-CTC5.0 criteria and RTOG/EORTC criteria.
Overall response rate | up to 5 years
  efficacy will be measured by PERCIST1.0 and RECIST1.1 criteria.

OTHER OUTCOMES:
Biomarkers | up to 5 years
  The correlation between the radiotherapy dose with biomarkers such as peripheral blood lymphocyte and EBV-DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Haihua Yang, MD, Principal Investigator — Taizhou Enze Medical Center Group
Locations (4):
- China (4):
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang
  - Taizhou Cancer Hospital, Taizhou, Zhejiang
  - Taizhou Enze Medical Center(Group) Enze Hospital, Taizhou, Zhejiang